CLINICAL TRIAL: NCT02867592
Title: Phase 2 Trial of XL184 (Cabozantinib) an Oral Small-Molecule Inhibitor of Multiple Kinases, in Children and Young Adults With Refractory Sarcomas, Wilms Tumor, and Other Rare Tumors
Brief Title: Cabozantinib-S-Malate in Treating Younger Patients With Recurrent, Refractory, or Newly Diagnosed Sarcomas, Wilms Tumor, or Other Rare Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01258; NCI-2016-01258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1622; ADVL1622 (Other: Children's Oncology Group); ADVL1622 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-08-15; First posted 2016-08-16 (Estimated); Results first posted 2022-11-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-06

CONDITIONS: Adrenal Cortical Carcinoma; Alveolar Soft Part Sarcoma; Central Nervous System Neoplasm; Childhood Clear Cell Sarcoma of Soft Tissue; Clear Cell Sarcoma of Soft Tissue; Ewing Sarcoma; Hepatoblastoma; Hepatocellular Carcinoma; Osteosarcoma; Recurrent Adrenal Cortical Carcinoma; Recurrent Alveolar Soft Part Sarcoma; Recurrent Clear Cell Sarcoma of Soft Tissue; Recurrent Ewing Sarcoma; Recurrent Hepatoblastoma; Recurrent Hepatocellular Carcinoma; Recurrent Kidney Wilms Tumor; Recurrent Malignant Solid Neoplasm; Recurrent Osteosarcoma; Recurrent Primary Malignant Central Nervous System Neoplasm; Recurrent Renal Cell Carcinoma; Recurrent Rhabdomyosarcoma; Recurrent Soft Tissue Sarcoma; Recurrent Thyroid Gland Medullary Carcinoma; Refractory Adrenal Cortical Carcinoma; Refractory Alveolar Soft Part Sarcoma; Refractory Clear Cell Sarcoma of Soft Tissue; Refractory Ewing Sarcoma; Refractory Hepatoblastoma; Refractory Hepatocellular Carcinoma; Refractory Malignant Solid Neoplasm; Refractory Osteosarcoma; Refractory Primary Central Nervous System Neoplasm; Refractory Primary Malignant Central Nervous System Neoplasm; Refractory Renal Cell Carcinoma; Refractory Rhabdomyosarcoma; Refractory Soft Tissue Sarcoma; Refractory Thyroid Gland Medullary Carcinoma; Refractory Wilms Tumor; Renal Cell Carcinoma; Rhabdomyosarcoma; Soft Tissue Sarcoma; Solid Neoplasm; Thyroid Gland Medullary Carcinoma; Wilms Tumor
MeSH Terms: conditions — Adrenocortical Carcinoma; Sarcoma, Alveolar Soft Part; Central Nervous System Neoplasms; Sarcoma, Clear Cell; Sarcoma, Ewing; Hepatoblastoma; Carcinoma, Hepatocellular; Osteosarcoma; Wilms Tumor; Carcinoma, Renal Cell; Rhabdomyosarcoma; Sarcoma; Carcinoma, Medullary | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib s-malate) (Experimental): Patients receive cabozantinib-s-malate orally (PO) on a continuous dosing schedule using a dosing nomogram on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib; Drug: Cabozantinib S-malate; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cabozantinib — Given PO
Drug: Cabozantinib S-malate — Given PO
  Note: Capsule formulation (Cometriq) not used in this trial.
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib-s-malate works in treating younger patients with sarcomas, Wilms tumor, or other rare tumors that have come back, do not respond to therapy, or are newly diagnosed. Cabozantinib-s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for tumor growth and tumor blood vessel growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate (complete response + partial response) of cabozantinib-s-malate (XL184) in children and young adults with Ewing sarcoma, rhabdomyosarcoma, non-rhabdomyosarcoma soft tissue sarcoma, and Wilms tumor.

II. To estimate whether XL184 therapy either improves the disease control rate at 4 months in patients with recurrent measurable osteosarcoma as compared to a historical Childrens Oncology Group (COG) experience or produces an objective response rate.

SECONDARY OBJECTIVES:

I. To further define XL184 related toxicities in pediatric, adolescent and young adult patients.

II. To further define XL184 pharmacokinetics in the pediatric and adolescent patients.

III. To estimate 1-year time to progression, progression free survival (PFS) and overall survival for each stratum, and if feasible to compare to historical controls.

EXPLORATORY OBJECTIVES:

I. To assess the effect of XL184 on patients' immune cell subsets. II. To obtain tumor tissue (snap frozen, formalin-fixed and paraffin-embedded [FFPE] blocks, or unstained slides) from diagnosis, recurrence, or both, for possible future studies.

OUTLINE:

Patients receive cabozantinib-s-malate orally (PO) on a continuous dosing schedule using a dosing nomogram on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 6 months for 1 year and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Upper age limit of =< 18 years of age for medullary thyroid carcinoma (MTC), renal cell carcinoma (RCC) and hepatocellular carcinoma (HCC) =< 30 years for all other diagnoses
* Patients must have a body surface area >= 0.35 m^2
* Patients must have recurrent or refractory disease, or newly diagnosed disease with no known curative therapy or therapy proven to prolong survival with an acceptable quality of life; patients must have had histologic verification of one of the malignancies listed below at original diagnosis or at relapse:

  * Ewing sarcoma
  * Rhabdomyosarcoma (RMS)
  * Non-rhabdomyosarcoma soft tissue sarcomas (STS) including microphthalmia transcription factor associated STS (alveolar soft part sarcoma [ASPS] and clear cell sarcoma [CCS])
  * Osteosarcoma
  * Wilms tumor
  * Rare tumors

    * Medullary thyroid carcinoma (MTC)
    * Renal cell carcinoma (RCC)
    * Hepatocellular carcinoma (HCC)
    * Hepatoblastoma
    * Adrenal coertex carcinoma
    * Pediatric solid tumors (including central nervous system [CNS] tumors) with known molecular alterations in the targets of XL184 (i.e., MET amplification, overexpression, activating mutation, MET translocation, MET exon skipping mutations, activating RET mutations, RET rearrangement, overexpression or activation of AXL); documentation of the alteration from a Clinical Laboratory Improvement Act (CLIA) certified laboratory will be required

      * Note: Documentation of any known tumor molecular alterations and RET mutation status for patients with MTC (germline) must be uploaded via the RAVE system
* Patients must have radiographically measurable disease; measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm)

  * Note: The following do NOT qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans)
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurement parameters noted above
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
* At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim
* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
* Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
* >= 2 weeks must have elapsed since local palliative radiation therapy (XRT) (small port); >= 6 weeks must have elapsed since treatment with therapeutic doses of M-Iodobenzylguanidine (MIBG); >= 3 months must have elapsed if prior craniospinal XRT was received, if >= 50% of the pelvis was irradiated, or if total-body irradiation (TBI) was received; >= 6 weeks must have elapsed if other substantial bone marrow irradiation was given

  * Subjects should not have any clinically relevant ongoing complications from prior radiation therapy (i.e., radiation esophagitis or other inflammation of the viscera)
* No evidence of active graft versus (vs.) host disease and >= 2 months must have elapsed since transplant
* Not previously received XL184 or another MET/HGF inhibitor (tivantinib or crizotinib); there are no limits on number of prior therapeutic regimens; patients who have been treated with prior VEGF pathway, or RET inhibitors (except XL184) may be eligible
* Peripheral absolute neutrophil count (ANC) >= 1000/uL for patients with solid tumors without bone marrow involvement
* Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment) for patients with solid tumors without bone marrow involvement
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) for patients with solid tumors without bone marrow involvement
* Peripheral absolute neutrophil count (ANC) >= 750/uL for patients with solid tumors and known bone marrow metastatic disease
* Platelet count >= 50,000/uL for patients with solid tumors and known bone marrow metastatic disease
* Hemoglobin >= 8.0 g/dL for patients with solid tumors and known bone marrow metastatic disease
* Transfusions are permitted to meet both the platelet and hemoglobin criteria for patients with known bone marrow metastatic disease; patients must not be known to be refractory to red blood cell or platelet transfusions
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 2 to < 6 years of age

    * Male and female: 0.8 (maximum serum creatinine [mg/dL])
  * 6 to < 10 years of age

    * Male and female: 1 (maximum serum creatinine [mg/dL])
  * 10 to < 13 years of age

    * Male and female: 1.2 (maximum serum creatinine [mg/dL])
  * 13 to < 16 years of age

    * Male 1.5 (maximum serum creatinine [mg/dL])
    * Female: 1.4 (maximum serum creatinine [mg/dL])
  * >= 16 years of age

    * Male: 1.7 (maximum serum creatinine [mg/dL])
    * Female: 1.4 (maximum serum creatinine [mg/dL])
* Urine protein: =< 30 mg/dl in urinalysis or =< 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hour (h) urine sample
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L (3 x ULN) (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2.8 g/dL
* No history of congenital prolonged corrected QT (QTc) syndrome, New York Heart Association (NYHA) class III or IV congestive heart failure (CHF)
* No clinically significant cardiac arrhythmias, stroke or myocardial infarction within 6 months prior to enrollment
* QTc =< 480 msec; Note: Patients with grade 1 prolonged QTc (450- 480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e., electrolytes, medications)
* Patients with a known seizure disorder who are receiving non-enzyme inducing anticonvulsants and have well-controlled seizures may be enrolled
* CNS toxicity =< grade 2 with the exception of decreased tendon reflex (DTR); any grade of DTR is eligible
* A blood pressure (BP) =< the 95th percentile for age, height, and gender for pediatric patients < 18 years old and =< 140/90 mmHg for patients >= 18 years old; patients should not be receiving medication for treatment of hypertension (except patients with Wilms tumor and RCC who may be eligible if on stable doses of no more than one anti-hypertensive medication with a baseline BP =< ULN for pediatric patients and =< 140/90 for adult patients); please note that 3 serial blood pressures should be obtained and averaged to determine baseline BP
* International normalized ratio (INR) =< 1.5
* Serum amylase =< 1.5 x ULN
* Serum lipase =< 1.5 x ULN

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use two methods of birth control- a medically accepted barrier method of contraceptive method (e.g., male or female condom) and a second effective method of birth control-during protocol therapy and for at least 4 months after the last dose of XL184; abstinence is an acceptable method of birth control
* Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment (14 days if pegfilgrastim)
* Patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Previous treatment with XL184 (cabozantinib) or another MET/HGF inhibitor (tivantinib, crizotinib)
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial
* Patients must not be receiving any of the following potent CYP3A4 inducers or inhibitors: erythromycin, clarithromycin, ketoconazole, azithromycin, itraconazole, grapefruit juice or St. John's wort
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin, direct thrombin, and Factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel) are prohibited

  * Note: Low-dose aspirin for cardioprotection (per local applicable guidelines) and low dose, low molecular weight heparins (LMWH) are permitted; anticoagulation with therapeutic doses of LMWH is allowed in subjects without radiographic evidence of brain metastasis, who are on a stable dose of LMWH for at least 6 weeks before first dose of study treatment, and who have had no complications from a thromboembolic event or the anticoagulation regimen
* Patients must not have received enzyme-inducing anticonvulsants within 14 days prior to enrollment
* Patients who are receiving drugs that prolong QTc are not eligible
* Patients who are unable to swallow intact tablets are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with active bleeding are not eligible; specifically, no clinically significant gastrointestinal (GI) bleeding, GI perforation, intra-abdominal abscess or fistula for 6 months prior to enrollment, no hemoptysis or other signs of pulmonary hemorrhage for 3 months prior to enrollment; patients with evidence of an acute intracranial or intratumoral hemorrhage on CT or MRI are not eligible (patients with evidence of resolving hemorrhage will be eligible); in patients with CNS tumors, an MRI with ECHO gradient sequences would be required to exclude presence of petechial hemorrhages
* Patients who have had or are planning to have the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, or open biopsy within 28 days prior to enrollment
  * Central line placement or subcutaneous port placement is not considered major surgery but must be placed at least 3 days prior to enrollment for external lines (e.g., Hickman or Broviac catheter, peripherally inserted central catheter [PICC]) and at least 7 days prior to enrollment for a subcutaneous port
  * Core biopsy within 7 days prior to enrollment
  * Fine needle aspirate within 7 days prior to enrollment
  * Surgical or other wounds must be adequately healed prior to enrollment
  * NOTE: For purposes of this study, bone marrow aspirate and biopsy are not considered surgical procedures and therefore are permitted within 14 days prior to start of protocol therapy
* Patients who have had significant traumatic injury within 28 days prior to enrollment are not eligible
* Patients with any medical or surgical conditions that would interfere with gastrointestinal absorption of the study drug are not eligible

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2026-06-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Srivandana Akshintala, Principal Investigator — Children's Oncology Group
Locations (142):
- United States (142):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Texas Tech University Health Sciences Center-El Paso, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Groups:
- Ewing's Sarcoma; Rhabdomyosarcoma; Non-Rhabdomyosarcoma Soft Tissue Sarcoma; Wilms Tumor; Rare Tumors; Osteosarcoma: Patients receive cabozantinib-s-malate (XL184), 40mg/m2/day orally (PO) on a continuous dosing schedule using a dosing nomogram on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
Started | 15 | 14 | 13 | 13 | 25 | 29
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 14 | 13 | 13 | 25 | 29
Not completed — Adverse Event | 3 | 0 | 2 | 1 | 1 | 5
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 8 | 10 | 8 | 8 | 12 | 17
Not completed — Physician Decision | 1 | 2 | 2 | 0 | 5 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 3 | 3
Not completed — Ineligible | 1 | 1 | 0 | 0 | 2 | 0
Not completed — No Treatment | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Still on Therapy | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Patient received concurrent anticancer or investigational therapy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Repeat Eligibility Studies (If Required) Are Outside The Parameters Required For Eligibility | 1 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma | Total
Number analyzed (Participants) | 15 | 14 | 13 | 13 | 25 | 29 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 8 | 11 | 22 | 17 | 71
  Between 18 and 65 years | 8 | 8 | 5 | 2 | 3 | 12 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 18.1 [7.3 to 26.8] | 19.3 [5.7 to 26.8] | 16.1 [10.1 to 26.3] | 14.1 [8.9 to 27.1] | 13.2 [5.6 to 19.5] | 16.8 [9.1 to 22.3] | 15.7 [5.6 to 27.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 10 | 15 | 10 | 53
  Male | 10 | 9 | 5 | 3 | 10 | 19 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 1 | 8 | 8 | 21
  Not Hispanic or Latino | 15 | 12 | 10 | 11 | 15 | 20 | 83
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 2 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 1 | 1 | 3 | 1 | 2 | 6 | 14
  White | 11 | 10 | 7 | 8 | 14 | 16 | 66
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 2 | 2 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Non-Osteosarcoma Strata)
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Response rates will be calculated as the percent of evaluable patients who are responders (Overall Best Response of Partial Response or Complete Response), and confidence intervals will be constructed accounting for the two-stage design.
Time Frame: Up to the first 6 cycles of therapy
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1622 protocol in non-osteosarcoma strata which were either statistical strata (Ewing's Sarcoma, Rhabdomyosarcoma, Non-Rhabdomyosarcoma Soft Tissue Sarcoma, and Rare Tumors) or accrued enough patients to be analyzed (Wilms Tumor). Data is limited for Rare tumors due to low accrual.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 23
Percentage of patients | 0 [0.0 to 24.71] | 0 [0.0 to 24.71] | 0 [0.0 to 24.71] | 0 [0.0 to 24.71] | 13.04 [2.78 to 33.59]

2. Primary Outcome: Objective Response (Osteosarcoma Stratum)
Description: Will be assessed by the Response Evaluation Criteria in Solid Tumors version 1.1 and Disease Control (see section 9.3.2 of the ADVL1622 Protocol). Response + Disease Control rate will be calculated as the percent of evaluable patients who are responders or who met the definition of disease control, and confidence intervals will be constructed accounting for the two-stage design.
Time Frame: Up to the first 6 cycles of therapy.
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1622 protocol in the osteosarcoma stratum.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Osteosarcoma
Number analyzed (Participants) | 29
Percentage of patients | 35.18 [20.16 to 48.27]

3. Secondary Outcome: Percentage of Participants With Adverse Events
Description: Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Will report the percentage of patients within each disease stratum who experienced a grade 3 or higher toxicity with attribution of possible, probable, or definite while on protocol therapy or within 30 days of the last dose of therapy
Time Frame: Up to 5 years (duration of protocol therapy plus 30 days after last dose of therapy)
Population: All patients who met the evaluable for toxicity criteria outlined in section 9.5 of the ADVL1622 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 23 | 29
Percentage of patients | 61.54 [31.58 to 86.14] | 38.46 [13.86 to 68.42] | 61.54 [31.58 to 86.14] | 38.46 [13.86 to 68.42] | 60.87 [38.54 to 80.29] | 68.97 [49.17 to 84.72]

4. Secondary Outcome: Pharmacokinetics (PK) Parameters of Cabozantinib S-malate: Cmax
Description: Day 1 PK peak concentration will be summarized by the mean and the standard deviation.
Time Frame: Prior to dose, 2, 4, 8 and 20-28 hours after dose on day 1
Population: All patients who consented to PK or were required to consent to PK and had enough samples to estimate the PK Parameter of interest.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- All Pharmacokinetic Patients: Patients receive cabozantinib-s-malate (XL184), 40mg/m2/day orally (PO) on a continuous dosing schedule using a dosing nomogram on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Pharmacokinetic Patients
Number analyzed (Participants) | 15
ng/mL | 567 (379.0)

5. Secondary Outcome: Pharmacokinetics (PK) Parameters of Cabozantinib S-malate: Tmax
Description: Day 1 PK time to peak concentration will be summarized by the mean and the standard deviation.
Time Frame: Prior to dose, 2, 4, 8 and 20-28 hours after dose on day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | All Pharmacokinetic Patients
Number analyzed (Participants) | 15
Hour | 2.9 (1.0)

6. Secondary Outcome: Pharmacokinetics (PK) Parameters of Cabozantinib S-malate: AUC
Description: Day 1 PK area under the curve will be summarized by the mean and the standard deviation.
Time Frame: Prior to dose, 2, 4, 8 and 20-28 hours after dose on day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | All Pharmacokinetic Patients
Number analyzed (Participants) | 16
hr*ng/mL | 7934 (4267.0)

7. Secondary Outcome: Pharmacokinetics (PK) Parameters of Cabozantinib S-malate: Accumulation
Description: PK accumulation will be summarized by the mean and the standard deviation.
Time Frame: Cycle 1, Day 1 (20-28 hours after dose) and Cycle 1, Day 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | All Pharmacokinetic Patients
Number analyzed (Participants) | 14
Ratio | 6.6 (6.0)

8. Secondary Outcome: Pharmacokinetics (PK) Parameters of Cabozantinib S-malate: Half-life
Description: PK half-life will be summarized by the mean and the standard deviation.
Time Frame: Cycle 1, Day 1 (20-28 hours after dose) and Cycle 1, Day 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | All Pharmacokinetic Patients
Number analyzed (Participants) | 14
Hour | 101 (100.1)

9. Secondary Outcome: Time to Progression (TTP)
Description: Percent of patients not yet progressed at 1 year as estimated by the Kaplan-Meier method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.1), as a >=20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Clinical progression was also counted as an event for this analysis.
Time Frame: Up to 1 year
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1622 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 23 | 29
Percentage of patients | 16.78 [2.67 to 41.51] | 0 [0 to 0] | 15.39 [2.48 to 38.78] | 23.08 [5.58 to 47.46] | 20.6 [5.89 to 41.42] | 21.25 [7.64 to 39.35]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: The 1-year Progression Free Survival will be estimated using Kaplan-Meier methodology. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECISTv1.1), as a >=20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 1 year
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1622 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 23 | 29
Percentage of patients | 15.39 [2.48 to 38.78] | 0 [0 to 0] | 15.39 [2.48 to 38.78] | 23.08 [5.58 to 47.46] | 13.04 [3.27 to 29.72] | 14.71 [4.66 to 30.19]

11. Secondary Outcome: Overall Survival (OS)
Description: The 1-year Overall Survival will be estimated using Kaplan-Meier methodology.
Time Frame: Up to 1 year
Population: All patients who met the evaluable for response criteria outlined in section 9.4 of the ADVL1622 protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 23 | 29
Percentage of patients | 53.85 [24.77 to 75.99] | 25 [6.01 to 50.48] | 74.59 [39.76 to 91.10] | 42.74 [15.90 to 67.50] | 34.78 [16.63 to 53.71] | 35.86 [18.96 to 53.13]

12. Other Pre Specified Outcome: Change in Immune Biomarkers
Description: The association between the host immune system and response to cabozantinib-s-malate will be assessed in an exploratory manner. each biomarker will be correlated with the clinical outcomes of objective response and progression free survival.
Time Frame: Baseline, day 1 (prior to dose) of cycles 2 and 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From start of treatment to 30 days after last dose, a median of 3.4 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Ewing's Sarcoma | Rhabdomyosarcoma | Non-Rhabdomyosarcoma Soft Tissue Sarcoma | Wilms Tumor | Rare Tumors | Osteosarcoma
All-Cause Mortality (participants affected / at risk) | 12/13 | 10/13 | 8/13 | 10/13 | 18/23 | 20/29
Serious Adverse Events (participants affected / at risk) | 6/13 | 2/13 | 4/13 | 6/13 | 10/23 | 8/29
Other Adverse Events (participants affected / at risk) | 5/13 | 7/13 | 7/13 | 7/13 | 13/23 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ewing's Sarcoma (N=13) | Rhabdomyosarcoma (N=13) | Non-Rhabdomyosarcoma Soft Tissue Sarcoma (N=13) | Wilms Tumor (N=13) | Rare Tumors (N=23) | Osteosarcoma (N=29)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Esophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 2 | 2 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ewing's Sarcoma (N=13) | Rhabdomyosarcoma (N=13) | Non-Rhabdomyosarcoma Soft Tissue Sarcoma (N=13) | Wilms Tumor (N=13) | Rare Tumors (N=23) | Osteosarcoma (N=29)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 3 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 3 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0 | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 1 | 2 | 4 | 1 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 0 | 1 | 4 | 2
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 2 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Serum amylase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 1
Weight loss (Investigations) | 0 | 1 | 2 | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
White blood cell decreased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT02867592/Prot_SAP_000.pdf